CLINICAL TRIAL: NCT01370343
Title: A Phase 1, Single-Dose, Open-Label, Crossover Study To Assess The Effect Of Cyclosporine On The Pharmacokinetics Of PF-04991532 In Healthy Adult Subjects
Brief Title: Single Dose Study Of The Effect Of Cyclosporine On The Pharmacokinetics Of PF-04991532 In Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2611010
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Healthy; Drug Interaction
MeSH Terms: interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04991532 alone (Experimental)
  Interventions: Drug: PF-04991532 alone
- PF-04991532 + cyclosporine (Experimental)
  Interventions: Drug: PF-04991532 + cyclosporine

INTERVENTIONS:
Drug: PF-04991532 alone — a single dose of 150 mg PF-04991532, fasted
  Arms: PF-04991532 alone
Drug: PF-04991532 + cyclosporine — a single dose of 150 mg PF-04991532 + a single dose of 600 mg cyclosporine, fasted
  Arms: PF-04991532 + cyclosporine

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of a single dose of PF-04991532 in healthy adult subjects with and without co-administration of cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests. Women must be of non childbearing potential as defined in Lifestyle Guidelines. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, sychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Subjects with clinically significant infections within the past 3 months (for example, those requiring hospitalization, or as judged by the Investigator), or evidence of any infection within the past 7 days.
* Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), on a single measurement [confirmed by a single repeat, if necessary] following at least 5 minutes of rest.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time profile (AUC) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hrs postdose
Max observed plasma concentration (Cmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hrs postdose

SECONDARY OUTCOMES:
Time of Cmax (Tmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hrs postdose
Terminal elimination half-life (t1/2) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hrs postdose
Total amount of unchanged drug excreted in the urine over 24 hours (Ae24) | 0-8, and 8-24hr postdose
Renal clearance (CLR) | 0-24hr
Total amount of unchanged drug excreted in the urine over 24 hours, expressed as percent of dose (Ae24(% excreted)) | 0-24hr

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611010&StudyName=Single%20Dose%20Study%20Of%20The%20Effect%20Of%20Cyclosporine%20On%20The%20Pharmacokinetics%20Of%20PF-04991532%20In%20Health%20Volunteers